CLINICAL TRIAL: NCT02078024
Title: Comparison of Ivermectin Alone With Albendazole (ALB) Plus Ivermectin (IVM) in Their Efficacy Against Onchocerciasis in the Volta Region, Ghana.
Brief Title: Efficacy of Ivermectin and Albendazole Against Onchocerciasis in the Volta Region, Ghana
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Christopher L. King, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: WU-10-205; CWRU-OCR-1 (Other: CWRU)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Onchocerciasis
Keywords: Onchocerciasis
MeSH Terms: conditions — Onchocerciasis | interventions — Intravital Microscopy; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Annual Ivermectin (Active Comparator): Ivermectin 200 µg/kg body weight given orally at 0, 12 and 24 months
  Interventions: Drug: IVM
- Biannual IVM 200 µg/kg plus ALB 800 mg (Experimental): IVM 200 µg/kg plus ALB 800 mg (regardless of weight) given at 0, 6, 12, 18, and 24 months.
  Interventions: Drug: IVM plus ALB
- Annual IVM 200 µg/kg plus ALB 800 mg (Experimental): IVM 200 µg/kg plus ALB 800 mg given at 0, 12 and 24 months; vitamin pills at given at 6 and 18 months.
  Interventions: Drug: IVM plus ALB
- Biannual IVM 200 µg/kg (Experimental): IVM 200 µg/kg given 0, 6, 12, 18, and 24 months.
  Interventions: Drug: IVM
- IVM 200 µg/kg plus ALB 400 mg (Experimental): IVM 200 µg/kg plus ALB 400 mg given at 0, 6, 12, 18, and 24 months.
  Interventions: Drug: IVM plus ALB

INTERVENTIONS:
Drug: IVM plus ALB
  Arms: Annual IVM 200 µg/kg plus ALB 800 mg; Biannual IVM 200 µg/kg plus ALB 800 mg; IVM 200 µg/kg plus ALB 400 mg
Drug: IVM
  Arms: Annual Ivermectin; Biannual IVM 200 µg/kg

SUMMARY:
We will examine whether a combination of Ivermectim (IVM) plus Albendazole (ALB) compared to IVM alone given annually, which is the current standard for mass drug administration (MDA), is more effective in sterilizing adult worms. We will also address whether IVM plus ALB given twice per year is superior to IVM given once per year or twice per year.

DETAILED DESCRIPTION:
We hypothesize that more effective combinations of dose schedules of existing antifilarial drugs for MDA against onchocerciasis could shorten the number of years needed to interrupt onchocerciasis transmission and eliminate this infectious disease in areas that previously had high disease rates. Improved treatments should also make it feasible to extend MDA into areas that are currently not being helped. These changes have the potential to completely change the game to make global elimination of onchocerciasis a feasible goal.

Participants will be randomized into 5 treatment arms with 75 subjects in each arm for a total of 375 and followed for 36 months after the initial treatment. The primary endpoint will be the percent fertile adult female worms in nodules removed 36 months after the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-60 years residing along the Kpassa in the Nkwanta North District of the Volta Region in Ghana
2. Two or more assessable onchocercal nodules
3. Skin microfilaria density ≥5mf/mg.

Exclusion Criteria:

1. Prior treatment with the antifilarial and/or anti-nematodal drugs diethylcarbamazine, suramin, ivermectin, albendazole, levamisole or >1week of treatment with doxycycline, within 12 months before planned test article administration.
2. Pregnant or breastfeeding women.
3. Low probability of residency in the area (based on subject's assessment) over the next 36 months.
4. Permanent disability, serious medical illnesses such as a stroke, advanced heart disease, uncontrolled diabetes, emphysema, etc. that prevents or impedes study participation and/or comprehension
5. Weight of <40kg suggesting malnourishment
6. Hemoglobin levels <7 gm/dL
7. aspartate aminotransferase, alanine aminotransferase, creatinine > 1.5 upper limit of normal.
8. Significant glycosuria or proteinuria (2+ or 3+ protein or glucose).
9. Known or suspected allergy to albendazole or ivermectin or other compounds related to these classes of medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 375 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
parasitologic efficacy | 36 months
  To compare the parasitologic efficacy, as measured by percent fertile adult female worms in nodules at 36 months after administration of annual doses of oral ivermectin alone versus ivermectin plus albendazole given annually or biannually in the treatment of subjects infected with Onchocerca volvolus

SECONDARY OUTCOMES:
additional measures of parasitologic efficacy | 0, 6, 12, 18, 24 and 36 months
  To compare additional measures of parasitologic efficacy of annual doses of oral ivermectin alone versus ivermectin plus albendazole given annually or biannually in the treatment of subjects infected with Onchocerca volvulus as measured by skin microfilaria levels at additional time points.
compare the percentage living versus dead female worms | 36 months
  To compare the percentage living versus dead female worms in nodules at 36 months following initiation of therapy of annual doses of oral ivermectin alone versus ivermectin plus albendazole given annually or biannually in the treatment of subjects infected with Onchocerca volvulus.
compare the number of nodules with intact microfilaria | 36 months
  To compare the number of nodules with intact microfilaria (Mf) at 36 months after administration annual doses of oral ivermectin alone versus ivermectin plus albendazole given annually or biannually in the treatment of subjects infected with Onchocerca volvulus.
assess different treatment regimens on Soil Transmitted Helminth infections | 0, 6, 12, 18, 24 and 36 months
  To assess different treatment regimens on Soil Transmitted Helminth (STH) infections based on presence and intensity of ova in stools.
determine if IVM plus ALB enhances immunological reactions | 0, 6, 12, 18, 24 and 36 months
  To determine if IVM plus ALB enhances immunological reactions to adult worms antigens, or release of circulating parasite antigens as potential biomarkers of drug efficacy.
determine if the host immune response facilitates killing or sterilizing adult worms and microfilariae | 0, 6, 12, 18, 24 and 36 months
  To determine if the host immune response facilitates killing or sterilizing adult worms and microfilariae. This can be accomplished by examining immune biomarkers prior to and following treatment using stored whole blood, and serum/plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L King, MD, PhD, Principal Investigator — Case Western Reserve University; James W Kazura, MD, Principal Investigator — Case Western Reserve University; Nicholas O Opoku, MBChB, MSc, Principal Investigator — Municipal Hospital, Hohoe, Ghana
Locations (1):
- Onchocerciasis Chemotherapy Research Centre, (OCRC) Municipal Hospital, Hohoe, Ghana